CLINICAL TRIAL: NCT04337489
Title: REmote MOniToring usE in Suspected Cases of COVID-19 (Coronavirus): REMOTE-COVID Trial
Brief Title: Remote Monitoring Use In Cases Of Suspected COVID-19 (Coronavirus)
Acronym: REMOTE-COVID
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: CW+ Charity (Other)
Responsible Party: Sponsor
Other Study IDs: REMOTE-COVID
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Coronavirus
Keywords: coronavirus; remote monitoring; deterioration; escalation
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: SensiumVitals wearable sensor — A waterproof, light, wearable sensor measuring vital signs (heart rate, respiratory rate, temperature) continuously.

SUMMARY:
The study aims to see if participant deterioration due to suspected coronavirus in a designated location (e.g. hotel) can be identified sooner by wearing the sensor. If sick patients can be identified early, participants are more likely to have better outcomes; the study believes that the sensor can help us do this. The sensor measures heart rate, respiratory rate and temperature every 2 minutes and this can be reviewed by the clinical team looking after the participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over.
* Able to provide written consent.

Exclusion Criteria:

* Any participants that withdraw their consent.
* A skin condition/reaction preventing wearing the wearable sensor.
* The presence of a permanent pacemaker or cardiac defibrillator.
* Any form of psychiatric disorder or a condition that, in the opinion of the investigator, may hinder communication with the research team.
* Inability to cooperate or communicate with the research team.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Returning traveller from a high-risk area into a London airport.
  * Have mild symptoms indicative of Covid-19
  * Unable to self-isolate
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Darzi, Prof, Principal Investigator — Institute of Global Health Innovation
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Result] Iqbal FM, Joshi M, Davies G, Khan S, Ashrafian H, Darzi A. The pilot, proof of concept REMOTE-COVID trial: remote monitoring use in suspected cases of COVID-19 (SARS-CoV 2). BMC Public Health. 2021 Apr 1;21(1):638. doi: 10.1186/s12889-021-10660-9. PMID 33794832
- [Derived] Iqbal FM, Joshi M, Davies G, Khan S, Ashrafian H, Darzi A. Design of the pilot, proof of concept REMOTE-COVID trial: remote monitoring use in suspected cases of COVID-19 (SARS-CoV-2). Pilot Feasibility Stud. 2021 Mar 5;7(1):62. doi: 10.1186/s40814-021-00804-4. PMID 33673868
- See also: Trial Protocol — https://pubmed.ncbi.nlm.nih.gov/33673868/
- See also: Published article — https://pubmed.ncbi.nlm.nih.gov/33794832/

RESULTS

PARTICIPANT FLOW:
Groups:
- Wearable Sensor: All participants had a wearable sensor applied
Period: Overall Study
Arm/Group | Wearable Sensor
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Wearable Sensor
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Deterioration Resulting in Healthcare Review
Description: Detection of clinical deterioration using wearable sensors resulting in healthcare review (e.g. GP telephone consultation)
Time Frame: 1 year
Measure: Number; unit: alerts generated
Arm/Group | Wearable Sensor
Number analyzed (Participants) | 14
alerts generated | 10

2. Secondary Outcome: Hospitalisation
Description: Deterioration resulting in hospitalisation
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Number of Individuals Hospitalised: All included participants
Arm/Group | Number of Individuals Hospitalised
Number analyzed (Participants) | 14
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: 0
Arm/Group | Wearable Sensor
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04337489/Prot_SAP_000.pdf
  • Informed Consent Form: Consent form (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT04337489/ICF_001.pdf